CLINICAL TRIAL: NCT04729712
Title: Ultrasound Guided Erector Spinae Plane (ESP) Catheter Versus Video-assisted Paravertebral Catheter Placement in Minimally Invasive Thoracic Surgery (MITS): Comparing Continuous Infusion Analgesic Techniques on Early Quality of Recovery, Respiratory Function, and Chronic Persistent Surgical Pain: A Multicentre, Randomised, Double-blind, Clinical Trial.
Brief Title: Efficacy of Ultrasound Guided ESP Vs Video-assisted PVB Catheter Placement in Minimally Invasive Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Aneurin Moorthy, Research Fellow in Anaesthesia and Perioperative Medicine, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESPvsPVB
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Regional Anesthesia Morbidity; Pain, Postoperative; Pain, Chronic
Keywords: Regional Anesthesia; Erector Spinae Block; Thoracic Paravertebral Block; Quality of Recovery; Chronic Persistent Surgical Pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Catheterization

STUDY DESIGN:
Intervention Model Description: This will be a multicentre, prospective, double-blinded, randomised controlled clinical trial. This study will take place between three level four academic hospitals in Co.Dublin, Ireland. One group will receive an Anaesthesiologist-administered, ultrasound guided erector spinae plane catheter and the other group will receive a surgeon-administered, video-assisted paravertebral catheter.
Who Masked: Participant, Outcomes Assessor
Masking Description: The erector spinae plane and paravertebral blocks with catheter insertion will be performed after induction of general anaesthesia and therefore participants will be blinded to which intervention they have had.
  The outcome assessors for this study will be unaware as to which group the participant will be randomised to and therefore they will be blinded to which intervention the participant had received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaesthesiologist-administered ultrasound guided Erector Spinae block with catheter insertion (Active Comparator): Patient's will be randomised to this arm of the study. This group will receive an erector spinae block with catheter insertion under ultrasound guidance under general anaesthesia. This regional anaesthesia procedure will be performed by an Anaesthesiologist with experience in performing this block.
  Interventions: Procedure: Anaesthesiologist-administered ultrasound guided Erector Spinae block with catheter insertion
- Surgeon-administered video-assisted Paravertebral block with catheter insertion (Experimental): Patient's will be randomised to this arm of the study. This group will receive a paravertebral block with catheter insertion under under thoracoscopic guidance. This regional anaesthesia procedure will be performed at the start of the operation by a surgeon with experience in performing this block.
  Interventions: Procedure: Surgeon-administered video-assisted Paravertebral block with catheter insertion

INTERVENTIONS:
Procedure: Anaesthesiologist-administered ultrasound guided Erector Spinae block with catheter insertion — Erector Spinae block: A bolus of 20 ml 0.375% Levobupivacaine will be administered into the erector spinae plane prior to surgical incision. A further bolus of 10 ml 0.25% Levobupivacaine will be given at skin closure if it has been greater than 1 hour after the first bolus of local anaesthetic medication. A continuous infusion of 0.125% Levobupivacaine will be commenced via the sited nerve catheter for postoperative analgesia. This will be started at 10 ml/hr and titrated to effect to a maximum rate of 15 ml/hr.
  Arms: Anaesthesiologist-administered ultrasound guided Erector Spinae block with catheter insertion
Procedure: Surgeon-administered video-assisted Paravertebral block with catheter insertion — Paravertebral block: A bolus of 20 ml 0.375% Levobupivacaine will be administered into the paravertebral space after the thoracoscopic ports have been sited. A further bolus of 10 ml 0.25% Levobupivacaine will be given at skin closure if it has been greater than 1 hour after the first bolus of local anaesthetic medication. A continuous infusion of 0.125% Levobupivacaine will be commenced via the sited nerve catheter for postoperative analgesia. This will be started at 10 ml/hr and titrated to effect to a maximum rate of 15 ml/hr.
  Arms: Surgeon-administered video-assisted Paravertebral block with catheter insertion

SUMMARY:
Minimally Invasive Thoracic Surgery (MITS) is a surgical method used to perform lung surgery through small incisions between the ribs and includes both Video-Assisted Thoracic Surgery (VATS) and Robotic assisted Thoracic Surgery (RATS). MITS can cause a significant amount of postoperative pain and if this is not adequately controlled, it can delay the patient's recovery and it may be a precipitating factor for the development of Chronic Persistent Surgical Pain (CPSP).

Regional anaesthesia is the use of nerve numbing medications known as local anaesthetics to block sensations of pain from a specific area of the body. For MITS, blocking pain arising from the chest wall/rib cage would improve the patient's recovery after the operation and overall patient satisfaction.

There have been significant advancements made in thoracic (chest wall) regional anaesthesia techniques. Ultimately, this involves injecting local anaesthetics around the nerves that supply the chest wall. A single injection of these medications will only have a maximum effect for up to 12 hours and often this is considerably less. To prolong the pain free benefit, a thin tube known as a catheter will be placed so that the local anaesthesia medication can be continuously given by a specific mechanical pump designed for this purpose. This mechanical pump will be located at the patient's bedside and can precisely deliver the medication in question at a rate between 10-15 ml/hr. This infusion of local anaesthesia medication will continue for 48 hours after the operation and will be monitored by the hospital's pain team.

The primary aim of this study is to compare the efficacy of two techniques for thoracic regional anaesthesia after this type of surgery. Participants will be randomly assigned (like tossing a coin) to receive either an Anaesthesiologist ultrasound guided Erector Spinae Plane Block (ESP) with catheter insertion or surgeon video-assisted Paravertebral block (PVB) with catheter insertion. Both these regional anaesthesia techniques are well established in clinical practice, but there is little evidence published comparing them for this type of surgery, in terms of quality of patient's short term (1-2 days) and longer-term (3 months) recovery.

DETAILED DESCRIPTION:
Erector Spinae Plane (ESP) block has emerged as a new regional anaesthesia technique which has had promising early results in attenuating severe acute pain associated with Minimal Invasive Thoracic Surgery (MITS). In a recent randomised control trial among MITS patients, single-shot ESP block improved Quality of Recovery score (QoR-15) and reduced overall complications at 24 hr compared with single-shot serratus anterior plane block (SAP).

Paravertebral block (PVB) has been widely used for analgesia after thoracic surgery for over two decades because it reduces postoperative pain and opioid requirements. When compared with systemic analgesia and alongside with epidural analgesia, it is considered the "gold standard" for thoracic regional analgesia techniques. Both ESP and PVB have usually been described as a single-shot technique. However, catheter techniques offer the prospect of flexibility and prolonged analgesia.

Placement of a thoracic PVB catheter can be achieved by an anatomical landmark or ultrasound technique. Ultrasound technique has a higher success rate and safer profile when compared to the landmark technique but is technically challenging. However, in MITS an opportunity arises for directly visualised placement of a PVB catheter by the surgeon under thoracoscopic guidance. Insertion of the PVB catheter and verification by the surgeon under direct vision could be a more reliable and safer method, but there are limited randomised controlled trials examining the efficacy of this technique. Also, there are limited clinical effectiveness trials on the catheter-based ESP analgesia technique using patient-centred outcomes. Furthermore, no study has evaluated the effect of acute analgesia over 24-48 hr with continuous regional nerve block on CPSP at 3 months after MITS.

Therefore, the investigators aim to complete a multicentre, prospective, double-blinded, randomised controlled clinical trial to test the hypothesis that Anaesthesiologist-administered, ultrasound guided ESP catheter analgesia is equivalent to surgeon-administered, video-assisted PVB catheter analgesia, in terms of early recovery (QoR-15), respiratory spirometric function at 24-48 hr, and CPSP at 3 months after MITS surgery.

Study setting: This study will take place between three level four academic hospitals in the Republic of Ireland (Mater Misericordiae Univeristy Hospital-MMUH, St Vincent's University Hospital-SVUH and St Jame's University Hospital-SJH).

Standard of care: Standard of care will be identical in both groups. The only difference will be that one group will receive an anaesthesiologist ultrasound guided placement of an erector spinae (ESP) catheter and the other will receive a surgeon video-assisted placement of a paravertebral block (PVB) catheter. Patients in both groups will be given a general anaesthetic as part of their care. All patients will be intubated with a double-lumen endotracheal tube and a radial arterial line will be sited for continuous haemodynamic monitoring. Venous access will be at the discretion of the consultant anaesthesiologist. The haemodynamic goal will be to maintain a systolic blood pressure within 20% of baseline and to avoid a heart rate greater than 100 beats per minute. Persistent hypertension and or tachycardia above this point will trigger an opioid (oxycodone, morphine or fentanyl) to be given intravenously. The frequency and dosage of this will be at the discretion of the anaesthesiology team.

Study intervention: Participants will be randomised into either the ESP or PVB group. No other forms of regional analgesia techniques (e.g. Intrathecal opioids, epidural analgesia, and subcutaneous infiltration of local anaesthetic) will be used during this trial.

Safety reporting: Any unexpected complications that may arise from this trial will be documented and reported to the principal investigator, surgical consultant and the relevant hospital patient safety board.

Sample size and justification: The primary outcome will be the QoR-15 score at 24 hours post operatively. The established minimum clinically important difference in QoR-15 is 8.0 and the SD of QoR-15 scores is typically between 10-16. [range of QoR score is 1-150]. We have chosen a SD of 12 to reflect our study population. Therefore, assuming Type I error = 0.05 and Type II error = 0.2 (80% power to detect this difference), then n=36 patients will be required in each group. We aim to enroll n=40 each group to allow for loss to follow up, missing data or withdrawal of consent.

Recruitment: Potential participants for this trial will be identified by a member of the surgical, anaesthetic or research team. A list of patients scheduled to have MITS will be made available the day before the procedure. These patients' electronic medical records will undergo a preliminary review to determine if they are potential candidates for this trial, i.e. if participants meet the inclusion criteria and have no exclusions.

The suitable patient will be approached the evening before surgery if available. Alternatively, patients will be approached on the ward on the morning of surgery and their suitability to participate in the trial will be confirmed. The purpose of the trial, peripheral nerve blocks (including benefits and risks) and method of follow up will be explained to the patient. A comprehensive and informative leaflet will be given to each patient and they will be afforded an adequate amount of time (minimum 10 mins) to study it. Participants will be informed that their participation in the study is entirely voluntary and they will have the opportunity to withdraw from the study at any time and this will not affect the quality of care they receive. Following this, participants will be offered an opportunity to ask any relevant questions and voice any potential concerns. If he/she professes an interest in participating in the trial written consent will be obtained. This process will be completed before transferring the patient to the theatre environment.

Study participants will be followed on Day 1 and Day 2 postoperatively for QoR-15 and spirometric score. A member of the research team will phone the patient at 3 months after the date of surgery and they will be asked to complete two questionnaires to assess for CPSP (BPI and SF-12)

Record Keeping: All patient data collected will be handled in accordance with European Union General Data Protection Regulations (EU 2016/679). Data will be initially collected manually and then transcribed onto Microsoft excel. Data collected from each hospital site will be stored securely in the Department of Anaesthesiology at the respective hospital, on a password-protected desktop computer stored in a locked office, such that only investigators assigned to data processing and analysis will have access to.

Statistical analysis: The collected raw data will be initially inspected for any errors, this includes but is not limited to double-entry errors, missing data and data that was incorrectly entered. Patients with missing or incorrect data will be excluded from the trial and this data will not be included in the final analysis. The data will be tested for normal distribution according to the Shapiro-Wilk test. Normally distributed data will be compared between the two groups using the unpaired student t-test and non-normal distributed data will be compared by using Mann-Whitney U test. All data will be summarised as mean + standard deviation and p value <0.05 will be considered statistically significant.

Financing and Insurance/Indemnity: Investigators in each hospital will be covered by the clinical indemnity scheme (CIS). No funding has been sought to conduct this clinical trial. Existing resources available to the investigators are sufficient to meet the aims of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants providing written informed consent
* American Society of Anesthesiologist grade 1-4
* Unilateral MITS (VATS and RATS) under general anaesthesia

Exclusion Criteria:

* Absence of written consent
* Unexpected conversion of MITS to open thoracotomy
* Contraindications to peripheral regional anaesthesia block: (Infection at local site, allergy to local anaesthesia medications, patient refusal, previous or existing neurological deficit, anticoagulated patients)
* Known dementia at time of MITS and inability to give informed consent
* Unexpected post-operative admission to ICU for continued ventilation
* History of opioid abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-15) score between Anaesthesiologist-administered ultrasound guided Erector Spinae block and Surgeon-administered video-assisted Paravertebral block at 24 hours postoperative. | 24 hours postoperative
  QoR-15 is a 15-parameter questionnaire which has been recommended as an optimum tool to evaluate overall patient recovery after surgery and this includes postoperative pain. Participants will complete this questionnaire at 24 hours after their surgery. It is scored between 0 and 150, where 150 indicates that the patient has had an excellent recovery.

SECONDARY OUTCOMES:
Chronic Persistent Surgical Pain (CPSP) after Minimally Invasive Thoracic Surgery (MITS) | 3 months postoperative
  Chronic Persistent Surgical Pain will be assessed at 3 months after MITS. This will be achieved by assessing the patient for chronic pain by using Brief Pain Inventory Short Form questionnaire. Brief Pain Inventory scale assess for quality of life and pain and its scale is measured between 0 - 10, where '0' indicates no interference with quality of life and no pain and '10' indicates severe interference with quality of life and severe pain. This assessment will be conducted by phone call between a member of the research team and the patient in question.
Chronic Persistent Surgical Pain (CPSP) after Minimally Invasive Thoracic Surgery (MITS) | 3 months postoperative
  Chronic Persistent Surgical Pain will be assessed at 3 months after MITS. This will be achieved by assessing the patient for chronic pain by using Short Form McGill questionnaire. Short Form McGill assess for neuropathic pain and its scale is measured between 0 - 100, where '0' indicates no neuropathic pain and '100' indicates severe neuropathic pain. This assessment will be conducted by phone call between a member of the research team and the patient in question.
Pulmonary Function Assessment | Preoperatively (day 0), postoperative day 1 and postoperative day 2
  Pulmonary function assessment will be evaluated preoperatively (day 0) before induction of general anesthesia (GA) and at postoperative day 1 and 2 using a bedside incentive spirometry. Maximum inspiration volume will be measured with the patient in the sitting position. A change in maximum inspiratory volumes between pre-operative and postoperative day 1 and 2 will be assessed.
Area Under the Curve (AUC) of Verbal Rating Score (VRS) for pain at rest and on deep inspiration versus time over 48 hours | 48 hours postoperative
  Verbal Rating scale is measured from 0 - 10, where '0' indicates no pain and '10' indicates severe pain.
Time of administration of first intravenous opioid | 48 hours postoperative
  The time (minutes) taken from immediately postoperative for the patient to receive first intravenous opioid.
Total 48 hours morphine consumption | 48 hours postoperative
  All patients will receive an opioid based patient control analgesia (PCA) as part of their postoperative analgesia plan. Total morphine consumption at 48 hours will be calculated.
Length of hospital stay | 1 month
  The length of in-patient stay (days).
Comprehensive Complication Index Calculator (CCI) | 1 month
  The CCI is calculated as the sum of all complications that are weighted for their severity. The final formula yields a continuous scale scale to rank the severity of any combination of complications from 0 to 100 in a single patient.
Documentation of adverse events | 48 hours postoperative
  This includes intra-operative haemodynamic changes, post-operative hypotension, nausea & vomiting, pruritis, block failure and block related complications.
Quality of Recovery (QoR-15) score between Anaesthesiologist-administered ultrasound guided Erector Spinae block and Surgeon-administered video-assisted Paravertebral block at 48 hours postoperative. | 48 hours postoperative
  QoR-15 is a 15-parameter questionnaire which has been recommended as an optimum tool to evaluate overall patient recovery after surgery and this includes postoperative pain. Participants will complete this questionnaire at 48 hours after their surgery. It is scored between 0 and 150, where 150 indicates that the patient has had an excellent recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Donal Buggy, MB Bch BAO, Principal Investigator — Professor of Anaesthesiology & Perioperative Medicine, Mater Misericordiae University Hospital,
Locations (2):
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - St Jame's University Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Yes
Individual Patient Data sharing will be supported with qualified external researchers and supporting clinical documents from eligible studies. All data provided will be coded and anonymised to respect the privacy of patients who have participated in the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years
Access Criteria: Publications, reports or query requests from future investigators.

REFERENCES:
- [Derived] Moorthy A, Ni Eochagain A, Dempsey E, Wall V, Marsh H, Murphy T, Fitzmaurice GJ, Naughton RA, Buggy DJ. Postoperative recovery with continuous erector spinae plane block or video-assisted paravertebral block after minimally invasive thoracic surgery: a prospective, randomised controlled trial. Br J Anaesth. 2023 Jan;130(1):e137-e147. doi: 10.1016/j.bja.2022.07.051. Epub 2022 Sep 13. PMID 36109206
- [Derived] Moorthy A, Eochagain AN, Dempsey E, Buggy D. Ultrasound-guided erector spinae plane catheter versus video-assisted paravertebral catheter placement in minimally invasive thoracic surgery: comparing continuous infusion analgesic techniques on early quality of recovery, respiratory function and chronic persistent surgical pain: study protocol for a double-blinded randomised controlled trial. Trials. 2021 Dec 28;22(1):965. doi: 10.1186/s13063-021-05863-9. PMID 34963493